CLINICAL TRIAL: NCT01510678
Title: The Effect of Three Different Dietary Messages on Dietary Intake and Health in Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 8721-B
Record Dates: First submitted 2012-01-05; First posted 2012-01-16 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Diet Quality
MeSH Terms: conditions — Obesity | interventions — Vegetables

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Decrease Condition (Experimental): In the Decrease Snack Foods condition participants will reduce intake of SFs (i.e., candy, cookies, cakes, ice cream, chips, nuts) to < 3 servings/week (for children aged 6 to 12 years, the solid fats and added sugar energy limit is 840 kcals/week and the DECREASE goal will help with meeting this limit). Children and parents will gradually work towards meeting these goals and self-monitor these behaviors.
  Interventions: Behavioral: Decrease Snack Foods
- Increase + Decrease Condition (Experimental): Families will be encouraged to increase fruits and vegetables and decrease snack foods.
  Interventions: Behavioral: Increase Fruits and Vegetables and Decrease Snack Foods
- Increase Condition (Experimental): A parent and child will be encouraged to increase fruits and vegetables. Children will be encouraged to consume 1 cup/day and 1.5 cups/day of whole fruit, and 1.5 cups/day and 2 cups/day of vegetables for children aged 6 to 8 years and 9 to 12 years, respectively. Children will gradually work towards these goals. Parents will also work towards F&V goals, with 2 cups/day of whole fruit and 2.5 cups/day of vegetables.
  Interventions: Behavioral: Increase Fruits and Vegetables

INTERVENTIONS:
Behavioral: Increase Fruits and Vegetables — Children will be encouraged to consume 1 cup/day and 1.5 cups/day of whole fruit, and 1.5 cups/day and 2 cups/day of vegetables for children aged 6 to 8 years and 9 to 12 years, respectively. Children will gradually work towards these goals. Parents will also work towards F&V goals, with 2 cups/day of whole fruit and 2.5 cups/day of vegetables. Both parent and child will self-monitor these behaviors. As one barrier to consuming F&Vs is perceived cost of these foods, information regarding lower-cost options for F&Vs will be included in the manual.
  Arms: Increase Condition
Behavioral: Decrease Snack Foods — This condition will reduce intake of SFs (i.e., candy, cookies, cakes, ice cream, chips, nuts) to < 3 servings/week (for children aged 6 to 12 years, the solid fats and added sugar energy limit is 840 kcals/week and the DECREASE goal will help with meeting this limit). Children and parents will gradually work towards meeting these goals and self-monitor these behaviors.
  Arms: Decrease Condition
Behavioral: Increase Fruits and Vegetables and Decrease Snack Foods — Will combine the goals of the increase and decrease conditions.
  Arms: Increase + Decrease Condition

SUMMARY:
Examine the effect of three different dietary messages on dietary intake and the health of parents and their children.

DETAILED DESCRIPTION:
The goal of this pilot study is to conduct a randomized controlled trial examining three dietary messages: increase fruits and vegetables [INCREASE], decrease energy-dense, non-nutrient dense snack foods [DECREASE], or increase fruits and vegetables plus decrease snack foods [INCREASE+DECREASE], within a 6-month, family-based obesity prevention intervention. Each condition will also focus on increasing family evening meals and physical activity. Primary hypotheses are: 1) INCREASE + DECREASE will consume a greater ratio of F&Vs:SFs than INCREASE and DECREASE at 6 months.

2)INCREASE + DECREASE will consume less energy than INCREASE and DECREASE at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 6-12 years
* BMI percentile > 5th and < 85th percentile for age and sex
* Have a parent aged > 21 years with a BMI > 25
* Have an overweight/obese parent willing to attend intervention meetings
* Parent and child speak and read English
* Not moving out of the metropolitan area during the course of the investigation

Exclusion Criteria:

* Reporting that the child and parent planning to participate have dietary restrictions related to fruit and vegetable intake
* Physical activity restrictions
* A parent reporting that she is pregnant, planning to become pregnant, or currently breastfeeding

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary intake | baseline and 6 months
  Changes in F&Vs, SFs, energy density, overall energy, and percent energy from fat intake, will be assessed by a three-day food record (two weekdays, one weekend day).

SECONDARY OUTCOMES:
Change in Anthropometrics | baseline and 6 months
  child and parent height, weight, BMI, and z-BMI
Change in Parent Feeding Styles | baseline and 6 months
  Includes 7 topics: perceived responsibility, perceived parent weight, perceived child weight, concern about child weight, restriction, pressure to eat, and monitoring.
Change in Parenting Styles | baseline and 6 months
  Assesses practices associated with different parenting styles
Change in Eating Pathology | baseline and 6 months
  Kids eating disorder survey and eating in the absence of hunger survey
Change in Physical Activity | baseline and 6 months
  Previous day physical activity recall- looks at 2 weekdays and 1 weekend day. For parents and children to complete
Change in Obesogenic Home Food Availability | baseline and 6 months
  self-report on foods that are available in the home.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, RD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - The University of Tennessee, Knoxville, Tennessee
  - Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee

REFERENCES:
- [Background] Birch LL, Ventura AK. Preventing childhood obesity: what works? Int J Obes (Lond). 2009 Apr;33 Suppl 1:S74-81. doi: 10.1038/ijo.2009.22. PMID 19363514
- [Background] Ebbeling CB, Ludwig DS. Pediatric obesity prevention initiatives: more questions than answers. Arch Pediatr Adolesc Med. 2010 Nov;164(11):1067-9. doi: 10.1001/archpediatrics.2010.186. No abstract available. PMID 21041601
- [Background] Davis MM, Gance-Cleveland B, Hassink S, Johnson R, Paradis G, Resnicow K. Recommendations for prevention of childhood obesity. Pediatrics. 2007 Dec;120 Suppl 4:S229-53. doi: 10.1542/peds.2007-2329E. PMID 18055653
- [Background] Cohen DA, Sturm R, Scott M, Farley TA, Bluthenthal R. Not enough fruit and vegetables or too many cookies, candies, salty snacks, and soft drinks? Public Health Rep. 2010 Jan-Feb;125(1):88-95. doi: 10.1177/003335491012500112. PMID 20402200
- [Background] Kral TV, Faith MS. Influences on child eating and weight development from a behavioral genetics perspective. J Pediatr Psychol. 2009 Jul;34(6):596-605. doi: 10.1093/jpepsy/jsn037. Epub 2008 Apr 10. PMID 18407923
- [Background] Carter FA, Bulik CM. Childhood obesity prevention programs: how do they affect eating pathology and other psychological measures? Psychosom Med. 2008 Apr;70(3):363-71. doi: 10.1097/PSY.0b013e318164f911. Epub 2008 Mar 31. PMID 18378876
- [Background] Golan M, Crow S. Parents are key players in the prevention and treatment of weight-related problems. Nutr Rev. 2004 Jan;62(1):39-50. doi: 10.1111/j.1753-4887.2004.tb00005.x. PMID 14995056
- [Background] Birch LL, Fisher JO. Development of eating behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):539-49. PMID 12224660
- [Background] Spear BA. Does dieting increase the risk for obesity and eating disorders? J Am Diet Assoc. 2006 Apr;106(4):523-5. doi: 10.1016/j.jada.2006.01.013. No abstract available. PMID 16567146
- [Background] Butryn ML, Wadden TA. Treatment of overweight in children and adolescents: does dieting increase the risk of eating disorders? Int J Eat Disord. 2005 May;37(4):285-93. doi: 10.1002/eat.20098. PMID 15856498
- [Background] Neumark-Sztainer D. Preventing obesity and eating disorders in adolescents: what can health care providers do? J Adolesc Health. 2009 Mar;44(3):206-13. doi: 10.1016/j.jadohealth.2008.11.005. PMID 19237105
- [Background] Epstein LH, Paluch RA, Consalvi A, Riordan K, Scholl T. Effects of manipulating sedentary behavior on physical activity and food intake. J Pediatr. 2002 Mar;140(3):334-9. doi: 10.1067/mpd.2002.122395. PMID 11953732
- [Background] Epstein LH, Roemmich JN, Paluch RA, Raynor HA. Influence of changes in sedentary behavior on energy and macronutrient intake in youth. Am J Clin Nutr. 2005 Feb;81(2):361-6. doi: 10.1093/ajcn.81.2.361. PMID 15699222
- [Background] Epstein LH, Roemmich JN, Paluch RA, Raynor HA. Physical activity as a substitute for sedentary behavior in youth. Ann Behav Med. 2005 Jun;29(3):200-9. doi: 10.1207/s15324796abm2903_6. PMID 15946114
- [Background] Epstein LH, Paluch RA, Beecher MD, Roemmich JN. Increasing healthy eating vs. reducing high energy-dense foods to treat pediatric obesity. Obesity (Silver Spring). 2008 Feb;16(2):318-26. doi: 10.1038/oby.2007.61. PMID 18239639
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Faith MS, Scanlon KS, Birch LL, Francis LA, Sherry B. Parent-child feeding strategies and their relationships to child eating and weight status. Obes Res. 2004 Nov;12(11):1711-22. doi: 10.1038/oby.2004.212. PMID 15601964
- [Background] Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, Flegal KM, Guo SS, Wei R, Mei Z, Curtin LR, Roche AF, Johnson CL. CDC growth charts: United States. Adv Data. 2000 Jun 8;(314):1-27. PMID 11183293
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Raynor HA. Evidence-based treatments for childhood obesity. In: Jelalian E, Steele R, eds. Handbook of Childhood and Adolescent Obesity. New York: Springer; 2008:201-220.
- [Background] Bronfenbrenner U. Ecological systems theory. Annals of Child Development. 1989;22:723-742.
- [Background] Tudor-Locke C, Johnson WD, Katzmarzyk PT. Accelerometer-determined steps per day in US children and youth. Med Sci Sports Exerc. 2010 Dec;42(12):2244-50. doi: 10.1249/MSS.0b013e3181e32d7f. PMID 20421837
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Ard JD, Fitzpatrick S, Desmond RA, Sutton BS, Pisu M, Allison DB, Franklin F, Baskin ML. The impact of cost on the availability of fruits and vegetables in the homes of schoolchildren in Birmingham, Alabama. Am J Public Health. 2007 Feb;97(2):367-72. doi: 10.2105/AJPH.2005.080655. Epub 2006 Nov 30. PMID 17138914
- [Background] Pinard CA, Davy BM, Estabrooks PA. Beverage intake in low-income parent-child dyads. Eat Behav. 2011 Dec;12(4):313-6. doi: 10.1016/j.eatbeh.2011.07.012. Epub 2011 Aug 1. PMID 22051366
- [Background] Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. Appetite. 2001 Jun;36(3):201-10. doi: 10.1006/appe.2001.0398. PMID 11358344
- [Background] Robinson CC, Mandelco B, Olsen SF, Hart CH. Authoritative, authoritarian and permissive parenting practices: Development of a new measure. Psychological Reports. 1995;77:819-830.
- [Background] Childress AC, Brewerton TD, Hodges EL, Jarrell MP. The Kids' Eating Disorders Survey (KEDS): a study of middle school students. J Am Acad Child Adolesc Psychiatry. 1993 Jul;32(4):843-50. doi: 10.1097/00004583-199307000-00021. PMID 8340308
- [Background] Fisher JO, Birch LL. Restricting access to foods and children's eating. Appetite. 1999 Jun;32(3):405-19. doi: 10.1006/appe.1999.0231. PMID 10336797
- [Background] Faith MS, Berkowitz RI, Stallings VA, Kerns J, Storey M, Stunkard AJ. Eating in the absence of hunger: a genetic marker for childhood obesity in prepubertal boys? Obesity (Silver Spring). 2006 Jan;14(1):131-8. doi: 10.1038/oby.2006.16. PMID 16493131
- [Background] Weston AT, Petosa R, Pate RR. Validation of an instrument for measurement of physical activity in youth. Med Sci Sports Exerc. 1997 Jan;29(1):138-43. doi: 10.1097/00005768-199701000-00020. PMID 9000167
- [Background] Fulkerson JA, Nelson MC, Lytle L, Moe S, Heitzler C, Pasch KE. The validation of a home food inventory. Int J Behav Nutr Phys Act. 2008 Nov 4;5:55. doi: 10.1186/1479-5868-5-55. PMID 18983668
- [Background] Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: Wiley & Sons; 1987.
- [Background] ACSM. ACSM Guidelines for Exercise Testing and Prescription 7th edition ed. Baltimore MD: Lippincott, Williams and Wilkins; 2006.
- [Background] Raynor HA, Osterholt KM, Hart CN, Jelalian E, Vivier P, Wing RR. Efficacy of U.S. paediatric obesity primary care guidelines: two randomized trials. Pediatr Obes. 2012 Feb;7(1):28-38. doi: 10.1111/j.2047-6310.2011.00005.x. Epub 2011 Dec 13. PMID 22434737
- [Background] Epstein LH, Gordy CC, Raynor HA, Beddome M, Kilanowski CK, Paluch R. Increasing fruit and vegetable intake and decreasing fat and sugar intake in families at risk for childhood obesity. Obes Res. 2001 Mar;9(3):171-8. doi: 10.1038/oby.2001.18. PMID 11323442